CLINICAL TRIAL: NCT04646850
Title: Long-term Treatment With the Ketogenic Diet in Epilepsy and Epilepsy-related Rare Diseases
Brief Title: Long-term Treatment With the Ketogenic Diet in Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anette Ramm-Pettersen, Head of Child Neurology, Oslo University Hospital
Other Study IDs: 18-14061
Record Dates: First submitted 2019-03-12; First posted 2020-11-30 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Epilepsy; GLUT1DS1; PDH Deficiency
Keywords: Ketogenic dieting
MeSH Terms: conditions — Epilepsy; Pyruvate Dehydrogenase Complex Deficiency Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Color duplex ultrasound of the carotid arteries — Examinations carried out according to the American Society of Echocardiography guidelines 25 using a Vivid 7 US instrumentation with a linear M12L probe (14 MHZ; General Electric).

SUMMARY:
This study will provide a comprehensive assessment of long-term treatment with the ketogenic diet, a medical diet with high fat and low carbohydrate intake, focusing on safety and cardiovascular implications. We will assess patients with epilepsy or one of two rare metabolic diseases; glucose transporter type 1 deficiency syndrome (GLUT1 DS) or pyruvate dehydrogenase complex deficiency (PDHD).

ELIGIBILITY:
Inclusion Criteria:

* Treatment with the ketogenic diet at the National Centre for Epilepsy (SSE) for 5 years or more
* Able to travel from The National Centre for Epilepsy - SSE (Sandvika) to Rikshospitalet (Gaustad) to perform procedures to investigate cardiovascular risk factors
* Willing to draw extra blood for research purposes
* Willing to sign informed consent and participate in the study in accordance with the study protocol
* Willing to sign informed consent for blood samples to be included in research biobank at the Department of Neurology, Oslo University Hospital

Exclusion Criteria:

* Non-compliance with the dietary treatment for 6 months or longer or more than once per month
* Not possible to communicate with parents in Norwegian or English without interpreter
* Patient not able to cooperate and lie still for about ten minutes during the carotid ultrasound examination
* Psychiatric/mental illness, alcohol or drug abuse or other factors making it impossible to pursue the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with the ketogenic diet (classical or modified) for epilepsy, GLUT1 deficiency or PDHD at The National Centre for Epilepsy - SSE for 5 years or longer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk after long-term treatment with the ketogenic diet | 2018-2022
  Color duplex ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Anette Ramm-Pettersen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway